CLINICAL TRIAL: NCT03293121
Title: Effect of Strength and Coordination Training on Biomechanics and Injury in New Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20010685
Record Dates: First submitted 2017-09-15; First posted 2017-09-26 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Injuries; Patellofemoral Pain Syndrome; Iliotibial Band Syndrome
Keywords: running related injuries
MeSH Terms: conditions — Wounds and Injuries; Patellofemoral Pain Syndrome; Iliotibial Band Syndrome | interventions — Walking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength and Coordination Training (Experimental): The strength and coordination group will perform a progression of exercises utilizing body weight and resistance bands as resistance. Exercises include squats, lunges, jumps etc. typical of a normal strength training program.
  Interventions: Behavioral: Strength and Coordination Training
- Walking (Active Comparator): The walking group will be instructed to walk 3x/week, progressing from 30 to 45 min over 8 weeks.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Strength and Coordination Training — Perform training exercises 3/week. Weeks 1-2: general strength (isolated muscle groups) Weeks 3-4: running-specific strength (multi-joint, upright) Weeks 5-6: power/coordination I (low amplitude/intensity) Weeks 7-8: power/coordination II (higher amplitude/intensity) Weeks 9-16: Run training. Each training session will start with a 10 minute strength & coordination warm up. Group will gradually progress from mixed run/walk for 20 minutes to a 40 minute run.
  Arms: Strength and Coordination Training
Behavioral: Walking — Perform training exercises 3/week. Weeks 1-2: 30 minute walk Weeks 3-4: 35 minute walk Weeks 5-6: 40 minute walk Weeks 7-8: 45 minute walk Weeks 9-16: Run training. Each training session will start with a 10 minute walking warm up. Group will gradually progress from mixed run/walk for 20 minutes to a 40 minute run.
  Arms: Walking

SUMMARY:
The investigators hypothesize that new runners participating in an 8 week strength and coordination training program prior to beginning to run will 1) display different coordination patterns , and 2) experience fewer injuries, compared to new runners who do not perform strength or coordination training prior to running.

DETAILED DESCRIPTION:
The study will investigate the effect of a sequenced training program - beginning with strength training, followed by running-specific coordination exercises, and finally a gradual introduction to running - on strength, coordination and injury incidence in a group of novice runners. he investigators hypothesize that runners who perform strength and coordination training prior to beginning to run will 1) demonstrate greater lower extremity strength, 2) demonstrate alters coordination patterns and 3) experience fewer injuries, when compared to a control group of novice runners who perform no physical preparation prior to a gradual introduction to running. The possible long-term benefits of this study include reduced burden of running-related injuries, increased participation in the sport of running, improved cardiovascular and metabolic health characteristics, and reduced incidence of disease such as cardiovascular events and cancer.

ELIGIBILITY:
Inclusion Criteria:

* No previous participation in running races
* Run less than 10km total in past year
* Able to run continuously (ie at least 5mph) for 5 min (so that biomechanical analysis of running form can be conducted)
* Female participants may not be pregnant
* Participants will be screened using the PARQ+ form, and Parmed-X form completed by a physician if necessary
* Cleared for physical activity through screening
* English-speaking

Exclusion Criteria:

* Previous (at any time of life) training of 3 or months of consistently running 3 or more days per week

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Running biomechanics | Change from week 0 to week 16
  Relative joint motions will be assessed continuously throughout the stride cycle using a vector coding technique.

SECONDARY OUTCOMES:
Running injury. | Measured in days over the 16 week training period.
  Time to first running related injury.

OTHER OUTCOMES:
Running performance | 16 weeks
  5km time trial at the end of 16 weeks training.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Finucane, PT, PhD, CEEAA, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States